CLINICAL TRIAL: NCT04944238
Title: Optimization of the Optical Constants of the PhysIOL ANKORIS Intraocular Lens
Brief Title: A-constant Optimization of a Toric Monofocal IOL
Status: Completed | Type: Observational
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PHY2014
Record Dates: First submitted 2021-06-18; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients implanted with Ankoris IOL: To assess the IOL stability, slitlamp photos of the consecutive 30 patients with respect to time will then be analysed with a 5% confidence interval.
  Interventions: Device: Ankoris

INTERVENTIONS:
Device: Ankoris — Implantations of test lens using standard phaco surgical technique, with aim for in-the-bag implantation.

SUMMARY:
The study is a prospective series study to determine the IOL constant of a hydrophilic toric monofocal intra-ocular lens (IOL)

DETAILED DESCRIPTION:
The study is a prospective series study with he principal objective to determine the IOL constant.

The secondary objectives of this study are to determine the rotational stability of the Ankoris intraocular lens and to measure the residual astigmatism after Ankoris IOL implantation with respect to the targeted astigmatism correction.

Although there may be no direct benefit to the subjects under study, the investigation will determined the optimized constant for accurate IOL power calculation and will assess the stability and efficacy of the toric optics: this would result in a benefit for the patient population. Since the material, the overall design of the IOL as well as the measuring procedure in this study is well tolerated in standard clinical practice and the IOL is readily available and CE-marked, the benefit/risk ratio appears acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 50 years old
* Age-related cataract
* Corneal astigmatisme >1 D
* Age 21 and older
* Visual Acuity > 0.05
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant.

Exclusion Criteria:

* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome, floppy iris syndrome, corneal pathologies
* Previous ocular surgery or trauma.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pseudophakic patients implanted with one of the two IOLs
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2019-06-11 (Actual)

PRIMARY OUTCOMES:
The principal objective of the study is to determine the IOL constant. | 1-2 hours
  IOL constant optimisation for PCI axial length measurement of Physiol Ankoris IOL.
The principal objective of the study is to determine the IOL constant. | 1 month
  IOL constant optimisation for PCI axial length measurement of Physiol Ankoris IOL.
The principal objective of the study is to determine the IOL constant. | 3 months
  IOL constant optimisation for PCI axial length measurement of Physiol Ankoris IOL.

SECONDARY OUTCOMES:
Rotational stability | 1-2 hours
  To measure the residual astigmatism after Ankoris IOL implantation with respect to the targeted astigmatism correction.
Rotational stability | 1 month
  To measure the residual astigmatism after Ankoris IOL implantation with respect to the targeted astigmatism correction.
Rotational stability | 3 months
  To measure the residual astigmatism after Ankoris IOL implantation with respect to the targeted astigmatism correction.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Sallet, MD, Principal Investigator — Private Eye Institue Aalst, Belgium
Locations (1):
- Guy Sallet, Aalst, Belgium

IPD SHARING:
Plan to Share IPD: No